CLINICAL TRIAL: NCT05544929
Title: A Phase I, Open-label, Multi-center Study of KFA115 as a Single Agent and in Combination With Pembrolizumab in Patients With Select Advanced Cancers
Brief Title: A Study of Safety and Efficacy of KFA115 Alone and in Combo With Pembrolizumab in Patients With Select Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKFA115A12101; 2022-502381-25 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2022-09-08; First posted 2022-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Cutaneous Melanoma; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Nasopharyngeal Carcinoma; Carcinoma, Thymic; Anal Cancer; Mesothelioma; Esophagogastric Cancer; High Microsatellite Instability Colorectal Carcinoma; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms
Keywords: Lung cancer; Non-small-cell lung cancer; NSCLC; Malignant Skin Cancer; Skin Cancer; Cutaneous melanoma; Renal cell carcinoma; RCC; Kidney cancer; Renal cancer; Clear cell carcinoma; Cancer of the ovaries; Female reproductive cancer; Ovarian carcinoma; Epithelial ovarian cancer; Nasopharyngeal Neoplasms; Nasopharyngeal carcinoma; NPC; Thymic carcinoma; Thymic tumor; Rectal cancer; Rectal neoplasms; Esophageal cancer; Cancer of throat; Colon cancer; Colorectal cancer; Bowel cancer; Cancer of the colon and rectum; High microsatellite instability colorectal carcinoma; CRC; MSI-H CRC; Advanced solid malignancies; Head and neck cancer; HNSCC; SCCHN; Squamous cell carcinoma of the head and neck; Cancer; Advanced cancer; NVP-KFA115; Triple Negative Breast Cancer; TNBC; Mesothelioma; Anal cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma; Carcinoma, Renal Cell; Carcinoma, Ovarian Epithelial; Nasopharyngeal Carcinoma; Thymoma; Anus Neoplasms; Mesothelioma; Squamous Cell Carcinoma of Head and Neck; Triple Negative Breast Neoplasms; Lung Neoplasms; Skin Neoplasms; Kidney Neoplasms; Adenocarcinoma, Clear Cell; Ovarian Neoplasms; Nasopharyngeal Neoplasms; Thymus Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Colonic Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Head and Neck Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single-agent KFA115 (Experimental): KFA115 monotherapy
  Interventions: Drug: KFA115
- KFA115 run-in (1 cycle) + pembrolizumab (Experimental): 1-cycle KFA115 run-in followed by addition of pembrolizumab
  Interventions: Drug: KFA115; Drug: pembrolizumab
- KFA115 + pembrolizumab (Experimental): KFA115 + pembrolizumab combination given concurrently
  Interventions: Drug: KFA115; Drug: pembrolizumab

INTERVENTIONS:
Drug: KFA115 — Immunomodulatory agent
  Other Names: NVP-KFA115
Drug: pembrolizumab — Anti-PD-1 antibody
  Other Names: Keytruda
  Arms: KFA115 + pembrolizumab; KFA115 run-in (1 cycle) + pembrolizumab

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of KFA115 and KFA115 in combination with pembrolizumab in patients with select advanced cancers, and to identify the maximum tolerated dose and/or recommended dose.

DETAILED DESCRIPTION:
This is a phase I, open-label, multi-center study of KFA115 as a single agent and in combination with pembrolizumab. The study consists of a dose escalation part, followed by dose expansion part(s) for single-agent KFA115 and KFA115 in combination with pembrolizumab. The escalation parts will characterize safety and tolerability. After the determination of the maximum tolerated dose (MTD) / recommended dose (RD), the dose expansion parts will assess the preliminary anti-tumor activity in defined patient populations and further assess the safety and tolerability at MTD/RD.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer with historic PD-L1 ≥ 1%, as determined locally using a clinically accepted assay. Patients must have experienced benefit from previous anti-PD(L)1-containing therapy for at least 4 months based on investigator-assessed disease stability or response prior to developing documented disease progression. Patients must have also received prior platinum-based chemotherapy, either in combination or in sequence with anti-PD-(L)1, unless patient was ineligible to receive such treatment.
* Renal cell carcinoma, clear cell histology, previously treated with anti-PD(L)1-containing therapy and a VEGF targeted therapy as monotherapy or in combination. Patients should have documented disease progression following anti-PD(L)1-containing therapy.
* Cutaneous melanoma, previously treated with anti-PD(L)1-containing therapy. Patients should have documented disease progression following anti-PD(L)1-containing therapy. Patients with BRAF V600-mutant melanoma must have also received prior therapy with a BRAF V600 inhibitor, with or without a MEK inhibitor.
* Ovarian cancer, high-grade serous histology, naïve to anti-PD(L)1 therapy, must have received one prior systemic therapy in platinum-resistant setting.
* Nasopharyngeal carcinoma, non-keratinizing locally advanced recurrent or metastatic. Depending on the study arm, patients may be naïve to anti-PD(L)1 therapy, or previously treated with platinum-based chemotherapy with or without anti-PD-(L)1.
* Locally advanced unresectable or metastatic triple negative breast cancer, ovarian cancer (high-grade serous histology), anal cancer (squamous), MSI-H CRC, esophagogastric cancer, mesothelioma, and HNSCC.
* Locally advanced unresectable or metastatic anal cancer (squamous), thymic carcinoma, MSI-H CRC, esophagogastric cancer, mesothelioma, and HNSCC, all naïve to anti-PD(L)1 therapy and for whom anti PD(L)1 therapy is not available.
* Triple negative breast cancer with historic PD-L1 CPS ≥ 1%, must have received at least one line of chemotherapy. In addition, these patients must have previously received sacituzumab govitecan, and in the case of a BRCA mutation a PARP inhibitor, if these treatments are locally approved and accessible to the patient.

Exclusion Criteria:

* Impaired cardiac function or clinically significant cardiac disease.
* Use of agents known to prolong the QT interval unless they can be permanently discontinued for the duration of study.
* History of severe hypersensitivity reactions to any ingredient of study drug(s) and other mAbs and/or their excipients.
* Active, known or suspected autoimmune disease. Patients with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur may be considered. Patients previously exposed to anti-PD-1/PD-L1 treatment who are adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.
* Any evidence of interstitial lung disease (ILD) or pneumonitis, or a prior history of ILD or non-infectious pneumonitis requiring high-dose glucocorticoids.
* Patients who discontinued prior anti-PD-(L)1 therapy due to an anti-PD-(L)1-related toxicity (applicable to the KFA115 in combination with pembrolizumab treatment arms).
* Patients with symptomatic peripheral neuropathy limiting instrumental activities of daily living.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-10-26 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose limiting toxicities (DLTs) during the DLT evaluation period of single-agent KFA115 (dose escalation only) | 28 days
  A DLT is defined as an adverse event or abnormal laboratory value that occurs during the DLT evaluation period where the relationship to study treatment cannot be ruled out, and is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications and meets the criteria defined in the study protocol
Incidence and severity of dose limiting toxicities (DLTs) during the DLT evaluation period of KFA115 in combination with pembrolizumab (dose escalation only) | 28 days
  A DLT is defined as an adverse event or abnormal laboratory value that occurs during the DLT evaluation period where the relationship to study treatment cannot be ruled out, and is not primarily related to disease, disease progression, intercurrent illness, or concomitant medications and meets the criteria defined in the study protocol
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 35 months
  Incidence and severity of adverse events and serious adverse events, including changes in laboratory values, vital signs, and electrocardiograms qualifying and reported as AEs
Frequency of dose interruptions, reductions | 35 months
  Number of dose interruptions of KFA115 and pembrolizumab, and number of dose reductions of KFA115
Dose intensity | 35 months
  Dose intensity of KFA115 and pembrolizumab is defined as the ratio of actual cumulative dose received and actual duration of exposure

SECONDARY OUTCOMES:
Best overall response (BOR) per RECIST v1.1 | 35 months
  BOR is defined as the best response recorded from the start of the treatment until disease progression/recurrence
Progression free survival (PFS) per RECIST v1.1 | 35 months
  PFS is defined as the time from date of start of treatment to the date of event defined as the first documented progression or death due to any cause
Duration of response (DOR) per RECIST v1.1 | 35 months
  DOR is defined as the time from the date of the first documented response (CR or PR) to the date of the first documented progression as per RECIST v1.1 or death due to underlying cancer
Time to progression (TTP) per RECIST v1.1 | 35 months
  TTP is defined as the time from date of start of treatment to the date of event defined as the first documented progression or death due to underlying cancer
Area under the concentration time curve (AUC) of KFA115 or pembrolizumab | During the first 168 days of treatment for single-agent KFA115 and 35 months for KFA115 in combination with pembrolizumab
  Area under the concentration time curve
Peak plasma or serum concentration (Cmax) of KFA115 or pembrolizumab | During the first 168 days of treatment for single-agent KFA115 and 35 months for KFA115 in combination with pembrolizumab
  The maximum (peak) observed plasma or serum drug concentration after single dose administration
Minimum plasma or serum concentration (Cmin) of KFA115 or pembrolizumab | During the first 168 days of treatment for single-agent KFA115 and 35 months for KFA115 in combination with pembrolizumab
  The minimum observed plasma or serum drug concentration reached during the time interval between two dose administrations
Time to reach peak plasma or serum concentration (Tmax) of KFA115 or pembrolizumab | During the first 168 days of treatment for single-agent KFA115 and 35 months for KFA115 in combination with pembrolizumab
  The time to reach maximum (peak) plasma or serum drug concentration after single dose administration
Elimination half-life (T1/2) of KFA115 or pembrolizumab | During the first 168 days of treatment for single-agent KFA115 and 35 months for KFA115 in combination with pembrolizumab
  The elimination half-life associated with the terminal slope of a semi logarithmic concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (5):
  - Massachusetts General Hospital ., Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - NYU School of Medicine, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - SCRI Oncology Partners, Nashville, Tennessee
- Novartis Investigative Site, Toronto, Ontario, Canada
- China (2):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Beijing
- Novartis Investigative Site, Lyon, France
- Germany (2):
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Essen
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No